CLINICAL TRIAL: NCT00898456
Title: Multidrug Resistance Protein Gene Polymorphisms in Acute Myeloid Leukemia. A CALGB Leukemia Tissue Bank Project
Brief Title: Multidrug Resistance Genes in Patients With Acute Myeloid Leukemia
Status: Active, not recruiting | Type: Observational
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: CALGB-20501; CALGB-20501; U10CA031946 (NIH); U10CA180821 (NIH); CDR0000514506 (Registry Identifier: NCI Physician Data Query)
Record Dates: First submitted 2009-05-09; First posted 2009-05-12 (Estimated); Last update posted 2023-08-18 (Actual); Status verified 2023-08

CONDITIONS: Leukemia
Keywords: adult acute myeloid leukemia; adult acute myeloid leukemia with 11q23 (MLL) abnormalities; adult acute myeloid leukemia with inv(16)(p13;q22); adult acute myeloid leukemia with t(16;16)(p13;q22); adult acute myeloid leukemia with t(8;21)(q22;q22); adult acute minimally differentiated myeloid leukemia (M0); adult acute myeloblastic leukemia without maturation (M1); adult acute myeloblastic leukemia with maturation (M2); adult acute myelomonocytic leukemia (M4); adult acute monoblastic leukemia (M5a); adult acute monocytic leukemia (M5b); adult erythroleukemia (M6a); adult pure erythroid leukemia (M6b); adult acute megakaryoblastic leukemia (M7); adult acute basophilic leukemia; adult acute eosinophilic leukemia
MeSH Terms: conditions — Leukemia; Leukemia, Myeloid, Acute; Congenital Abnormalities; Leukemia, Myelomonocytic, Acute; Leukemia, Monocytic, Acute; Leukemia, Erythroblastic, Acute; Leukemia, Megakaryoblastic, Acute; Leukemia, Basophilic, Acute; Leukemia, Eosinophilic, Acute | interventions — Gene Expression Profiling; Genetic Testing; Amplified Fragment Length Polymorphism Analysis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Group 1: Leukemia blast cells obtained from bone marrow aspirate or peripheral blood at diagnosis are used to study polymorphisms and haplotypes of ATP-binding cassette (ABC) B1, ABCC1, ABCG2, and other candidate genes. Multidrug resistance (MDR) protein expression and function are also analyzed using leukemia blast cells from patients enrolled on CALGB-9760.
  Interventions: Genetic: gene expression analysis; Genetic: molecular genetic technique; Genetic: polymorphism analysis; Genetic: protein expression analysis; Other: diagnostic laboratory biomarker analysis

INTERVENTIONS:
Genetic: gene expression analysis
Genetic: molecular genetic technique
Genetic: polymorphism analysis
Genetic: protein expression analysis
Other: diagnostic laboratory biomarker analysis

SUMMARY:
This research trial studies multidrug resistance genes in patients with acute myeloid leukemia. Studying samples of bone marrow or blood from patients with cancer in the laboratory may help doctors learn more about changes that may occur in deoxyribonucleic acid (DNA) and identify biomarkers related to cancer. It may also help doctors learn more about drug resistance and how patients respond to treatment.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To investigate the association of common single nucleotide polymorphisms (SNPs) and haplotypes of the three multidrug resistance (MDR) genes with treatment outcome in the clinical studies.

II. To assess the effect of ATP-binding cassette (ABC) B1, ABCC1, and ABCG2 polymorphisms and haplotypes on treatment outcome in younger patients enrolled on Cancer and Leukemia Group B (CALGB) 9621 and 19808.

III. To assess the effect of ABCB1, ABCC1, and ABCG2 polymorphisms and haplotypes on treatment outcome in older patients enrolled on CALGB 9720.

SECONDARY OBJECTIVES:

I. To test the hypothesis that ABCB1, ABCC1, and ABCG2 polymorphisms and haplotypes are associated with phosphoglycolate phosphatase (Pgp), multidrug resistance protein 1 (MRP-1), and ATP-binding cassette, sub-family G (WHITE), member 2 (Junior blood group) (BCRP) function and expression in pre-treatment blasts from acute myeloid leukemia (AML) patients.

II. To assess the effect of ABCB1, ABCC1, and ABCG2 polymorphisms and haplotypes on PGP, MRP-1, and BCRP function through CALGB 9760 in younger patients enrolled on CALGB 9621 and 19808.

III. To assess the effect of ABCB1, ABCC1, and ABCG2 polymorphisms and haplotypes on PGP, MRP-1, and BCRP function through CALGB 9760 in older patients from CALGB 9720.

IV. To conduct an exploratory analysis of the association of additional candidate genes relevant to etoposide, cytarabine, and daunorubicin with chemotherapy response and toxicity.

OUTLINE:

Leukemia blast cells obtained from bone marrow aspirate or peripheral blood at diagnosis are used to study polymorphisms and haplotypes of ATP-binding cassette (ABC) B1, ABCC1, ABCG2, and other candidate genes. Multidrug resistance (MDR) protein expression and function are also analyzed using leukemia blast cells from patients enrolled on CALGB-9760.

PROJECTED ACCRUAL: Tissue samples from over 600 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of acute myeloid leukemia
* Treated on protocols CALGB-9621, CALGB-9720, or CALGB-19808
* Registered on the mandatory companion Leukemia Tissue Bank Protocol CALGB-9665

  * Registration on another companion trial, CALGB-9760, (Multidrug Resistance Studies in Acute Leukemia) allowed

PATIENT CHARACTERISTICS:

* Not specified

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with acute myeloid leukemia enrolled on CALGB-9621, CALGB-9720, or CALGB-19808
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2006-10; Primary Completion 2100-01 (Estimated)

PRIMARY OUTCOMES:
Correlation of common single nucleotide polymorphisms (SNPs) and haplotypes of the 3 multidrug resistance genes (P-glycoprotein [Pgp], multidrug resistance-associated protein (MRP-1) and breast cancer resistance protein [BCRP]) with treatment outcome | Baseline
Effect of ATP-binding cassette (ABC) B1, ABCC1, and ABCG2 polymorphisms on treatment outcome | Baseline

SECONDARY OUTCOMES:
Association of ABCB1, ABCC1, and ABCG2 polymorphisms and haplotypes with Pgp, MRP-1, and BCRP function and expression in pre-treatment blasts | Baseline
Effect of ABCB1, ABCC1, and ABCG2 polymorphisms and haplotypes on Pgp, MRP-1, and BCRP function | Baseline
Association of additional candidate genes relevant to etoposide, cytarabine, and daunorubicin with chemotherapy response and toxicity | Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Maria R. Baer, MD, Study Chair — University of Maryland Greenebaum Cancer Center
Locations (1):
- Fort Wayne Medical Oncology and Hematology, Fort Wayne, Indiana, United States